CLINICAL TRIAL: NCT07235410
Title: Deep Learning-Based Multidimensional Body Composition Mapping for Predicting Clinical Outcomes in Hepatocellular Carcinoma Patients Undergoing TACE
Brief Title: Deep Learning-Based Multidimensional Body Composition Mapping for Outcome Prediction in HCC Patients Undergoing TACE
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lian Yang, Archiater, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: [2025](1186)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is a common liver cancer, and many patients cannot receive surgery. For these patients, transarterial chemoembolization (TACE) is an important treatment. However, patients often respond differently to TACE, and it is difficult to predict who will benefit most. This study uses deep learning to automatically analyze routine CT images taken before TACE. By measuring body composition features, such as the size and condition of different abdominal organs and tissues, we aim to better understand patients' overall health status and treatment tolerance. The goal is to develop a prediction model that can help doctors estimate survival and treatment outcomes more accurately. This may assist in making more personalized treatment decisions and improving patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with "Hepatocellular Carcinoma" from January 1, 2018 to May 31, 2024;
2. Age > 18 years old.

Exclusion Criteria:

1. Poor image quality;
2. Loss of follow-up;
3. Presence of another type of malignant tumor other than liver cancer;
4. Incomplete medical records.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
OS | After the TACE procedure until May 1, 2025

SECONDARY OUTCOMES:
PFS | After the TACE procedure until May 1, 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No